CLINICAL TRIAL: NCT05238558
Title: A Phase I Study of FMPV-1 in Healthy Male Subjects to Assess Safety and Immune Response
Brief Title: Safety and Immune Response to FMPV-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hubro Therapeutics AS (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMPV-1-01; QSC204718 (Other: Quotient)
Record Dates: First submitted 2022-01-26; First posted 2022-02-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer
Keywords: FMPV-1; Cancer-specific vaccine; Neoantigen; GM-CSF adjuvant
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMPV-1 vaccination (Experimental): GM-CSF (0.03 mg) + FMPV-1 (0.15 mg/injection: low dose) administered as 2 separate intradermal injections.
  Total of 8 administrations intradermally; GM-CSF + FMPV-1 on 5 separate occasions and FMPV-1 (without GM-CSF) on 3 occasions for the DTH skin reactivity assessment.
  Interventions: Biological: FMPV-1; Biological: GM-CSF (as adjuvant)

INTERVENTIONS:
Biological: FMPV-1 — Intradermal administration
Biological: GM-CSF (as adjuvant) — Intradermal administration

SUMMARY:
This is a single centre, open-label, non-randomized, Phase I study assessing safety and immune response of FMPV-1 in healthy male subjects.

DETAILED DESCRIPTION:
To date, there is no clinical experience with FMPV-1. This is the first clinical study with FMPV-1 in healthy volunteers to assess the safety and immunogenicity of FMPV-1 in man. The study population will include 16 healthy males in 2 cohorts (8 per cohort) to ensure data in a minimum of 14 subjects.

Up to two dose levels of FMPV-1 in conjunction with the adjuvant granulocyte macrophage colony stimulating factor (GM-CSF) will be assessed - the dose in Cohort 2 will depend on the safety and specific delayed type hypersensitivity (DTH) response data from Cohort 1. Each cohort will follow the same study design. Following preliminary screening procedures, subjects will be admitted in the morning on the day before initial dosing (Day -1). In Cohorts 1 and 2, subjects will receive FMPV-1 15 ± 5 min after GM-CSF on Days 1, 8, 15, 29 and 43 as an intradermal injection into the back of the upper arm. In Cohort 1, 8 subjects will receive GM-CSF (0.03 mg) + FMPV-1 (0.15 mg/injection: low dose) administered as 2 separate intradermal injections. In Cohort 2, 8 subjects will receive GM-CSF (0.03 mg) + FMPV-1 (either 0.15 or 0.3 mg/injection - dependent on Cohort 1 data) administered as 2 separate intradermal injections.

Sentinel dosing will be applied for both cohorts if different doses are used; if the same dose is to be used in both cohorts, sentinel dosing will not be applied in Cohort 2.

Adverse events and laboratory assessments will be the endpoints to assess the safety of GM-CSF/FMPV-1 vaccination. FMPV-1 specific DTH responses and FMPV-1-specific proliferative T-cell responses will be the endpoints to assess the FMPV-1 specific immune response. Subjects will receive a total of 8 administrations intradermally: GM-CSF + FMPV-1 on 5 separate occasions and FMPV-1 (without GM-CSF) on 3 occasions for the DTH skin reactivity assessment. The main part of the study will last for approximately 16 weeks, including screening, and subjects will return for follow-up visits after 6 months and 12 months. The overall estimated time from screening until the final follow-up visit is approximately 12 months. All adverse reactions will be collected until early withdrawal or discharge from the study after the 12-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Aged 18 to 55 years inclusive at the time of signing informed consent
3. Body mass index (BMI) of 18.0 to 32.0 kg/m2 as measured at screening
4. Must provide written informed consent
5. Must agree to adhere to the contraception requirements: male subjects who are sexually active with a partner of childbearing potential must use a condom plus an approved method of highly effective contraception from the time of informed consent until 90 days (one cycle of spermatogenesis) after last vaccine administration.

Exclusion Criteria:

1. Subjects who have received any investigational medicinal product in a clinical research study within the 90 days prior to Day 1 or within less than 5 elimination half-lives prior to Day 1, whichever is longer
2. Subjects who are, or are immediate family members of, a study site or sponsor employee
3. Subjects who have previously been administered investigational medicinal product in this study.
4. Evidence of current SARS-CoV-2 infection
5. History of any drug or alcohol abuse in the past 2 years
6. Regular alcohol consumption defined as >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
7. A confirmed positive alcohol breath test at screening or admission
8. Current smokers and those who have smoked within the last 6 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
9. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 6 months
10. Subjects with pregnant or lactating partners
11. Clinically significant abnormal clinical chemistry, haematology, coagulation or urinalysis as judged by the investigator. Subjects with Gilbert's Syndrome are not allowed.
12. Confirmed positive drugs of abuse test result
13. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results
14. History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
15. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
16. Presence or history of a clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
17. Subjects currently receiving any agent with a known effect on the immune system within 90 days before first investigational medicinal product administration
18. Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood
19. Subjects who are taking, or have taken, any prescribed or over-the-counter medications, herbal remedies or antihistamines (other than vitamin supplements and/or up to 4 g of paracetamol per day) in the 7 days before investigational medicinal product administration
20. Subjects who have had a vaccine (including COVID-19 vaccine) within 28 days before first dose
21. Subjects with tattoos or scars on the arms which may interfere with injection site assessments, as determined by the investigator or delegate at screening
22. Subjects with any other illnesses or medical conditions such as, but not limited to:

    * Any infection that requires systemic treatment (any grade)
    * Cardiac failure (any grade)
    * Systemic and gastrointestinal inflammatory conditions
    * Bone marrow dysplasia
    * History of auto-immune disease
    * History of adverse reactions to any vaccines
    * History of adverse reactions to GM-CSF
23. Subjects with any other malignancies within the last 3 years (except for adequately treated carcinoma of the cervix or basal or squamous cell skin cancer)
24. Subjects planning to receive a yellow fever or other live (attenuated) vaccine during the course of study
25. Subject has a first degree relative with a haematological malignancy
26. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Delayed Type Hypersensitivity Skin Reactivity Test | 45 days
  DTH test performed on Days 3, 29 and 43 with response assessment on Days 8, 31 and 45. A positive DTH response will be recorded if the area of the skin reaction (redness and/or induration) at the injection site has an average diameter ≥5 mm 48 h after injection.
Proliferative T-cell Responses | 12 months
  Whole Blood Samples for Proliferative T-cell Responses taken on Days 1, 45, 57±1, 80±3, 6-month and 12-month follow-ups. Samples will be processed to isolate PBMCs for T-cell receptor analysis.
Summary of Adverse Events | 12 months
  An AE is any untoward medical occurrence in a subject that occurs either before dosing (referred to as a pre-dose AE) or once a medicinal product has been administered, including occurrences which are not necessarily caused by or related to that product. AEs will be monitored from the time the subject signs the ICF until after the 12-month follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nand Singh, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Inderberg EM, Singh N, Miller R, Arbe-Barnes S, Eriksen HK, Lversen B, Juul HV, Eriksen JA, Handeland KR. Generation of frameshift-mutated TGFbetaR2-specific T cells in healthy subjects following administration with cancer vaccine candidate FMPV-1/GM-CSF in a phase 1 study. Cancer Immunol Immunother. 2025 Feb 25;74(4):115. doi: 10.1007/s00262-025-03969-6. PMID 39998682